CLINICAL TRIAL: NCT02939807
Title: A Phase II Study of ABC294640 in Patients With Advanced Hepatocellular Carcinoma Who Have Progressed on Sorafenib
Brief Title: A Phase II Study of ABC294640 as Monotherapy in Patients With Advanced Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study is being rewritten for different disease population
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Apogee Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102418; ABC-106 (Other: Medical University of South Carolina); 1P01CA203628-01 (NIH)
Record Dates: First submitted 2016-10-12; First posted 2016-10-20 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Yeliva™; hepatocellular carcinoma; ABC294640; hepatic neoplasms; liver neoplasms; hepatic cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- advanced HCC, tumor progression with sorafenib (Experimental): Patients with advanced HCC who have experienced tumor progression with sorafenib will receive ABC294640.
  Interventions: Drug: ABC294640

INTERVENTIONS:
Drug: ABC294640 — ABC294640 500 mg orally twice daily (approximately 12 hours apart) continuously.
  ABC294640 will be dosed under fasting conditions (at least 1 hour before or 2 hours after eating). A cycle is defined as 28 days.
  Other Names: YelivaTM

SUMMARY:
This is a Phase II study of single agent ABC294640. Patients with advanced hepatocellular carcinoma (HCC) who have experienced tumor progression or unacceptable toxicity on single agent sorafenib will receive ABC294640 500 mg by mouth twice a day continuously. Patients will continue on study drug until the development of progressive disease per modified RECIST, intolerable toxicity, withdrawal of patient consent or other event as outlined in patient discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have advanced hepatocellular carcinoma; fibrolamellar HCC is not allowed. Hepatocellular carcinoma will be confirmed by at least one of the following:

   1. Tissue diagnosis
   2. The presence of one or more liver lesions measuring 2 cm in longest diameter, showing characteristic arterial enhancement and venous washout using arterial-phase contrast enhanced imaging, and a clinical history of cirrhosis.(1)
2. Voluntary signed and dated institutional review board (IRB) approved informed consent form in accordance with regulatory and institutional guidelines.
3. Documented progression or intolerance to sorafenib as determined by the enrolling investigator:
4. Patient must have at least one measurable untreated lesion as per modified RECIST criteria. Measurable disease may include extrahepatic lesions. Abdominal imaging should employ a "liver protocol" image capture technique. The following are not considered measurable lesions: bone lesions, ascites, and pleural effusions. Prior RFA, PEI, or TACE of non-target lesions is allowed.
5. Time interval for last local therapy (radiofrequency ablation, percutaneous ethanol injection, radiotherapy, transarterial chemoembolization) more than 4 weeks prior to registration.
6. Life expectancy of at least 12 weeks.
7. 18 years of age or older.
8. ECOG performance status of 0-2.
9. Child-Pugh Cirrhotic Status A or B with a score of 7.
10. Acceptable liver function:

    1. Bilirubin ≤ 3 times upper limit of normal (CTCAE Grade 2 baseline)
    2. AST (SGOT), ALT (SGPT) 3 x ULN (CTCAE Grade 1 baseline)
11. Acceptable kidney function:

    a. Serum creatinine ≤ 1.5 XULN (CTCAE Grade 1 baseline)
12. Acceptable hematologic status:

    1. Absolute neutrophil count 1000 cells/mm3
    2. Platelet count 75,000 (plt/mm3), (CTCAE Grade 1 baseline)
    3. Hemoglobin 9 g/dL.
13. Acceptable blood sugar control

    a. Fasting glucose < 160 mg/dL (CTCAE grade 1 baseline)
14. Urinalysis: No clinically significant abnormalities.
15. INR < 1.7
16. As determined by the treating investigator, the patient must have well-controlled blood pressure, defined as systolic blood pressure <150mmHg and/or diastolic blood pressure <100 mmHg for the majority of measurements.
17. A negative pregnancy test (only for WOCBP).
18. Willingness to use effective contraceptive methods during the study. If patient is female (or female partner of male subject), must be either not of childbearing potential (defined as postmenopausal for ≥ 1 year or surgically sterile) or is practicing two forms of contraception. Sexually active male participants must agree to use a physical barrier method (male latex rubber condom with or without spermicide).

Exclusion Criteria:

1. New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG.
2. Underlying psychiatric disorder requiring hospitalization within the last two years or a HADS score of 11 or more.
3. Clinically significant neurological disorder (Parkinson's disease, dementia, multiple sclerosis), as determined by the enrolling investigator
4. Active, uncontrolled bacterial, viral or fungal infection, requiring systemic therapy.
5. Pregnant or nursing women. NOTE: Women of childbearing potential and men must agree to use adequate contraception or abstinence prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
6. Treatment with radiation therapy, surgery, or investigational therapy within one month prior to registration.
7. More than two lines of prior systemic therapy for HCC
8. Unwillingness or inability to comply with procedures required in this protocol.
9. Known infection with HIV.
10. Hepatitis C on protease therapy.
11. Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator.
12. Patients who are receiving drugs that are sensitive substrates of CYP450 1A2, 3A4, 2C9, 2C19 or 2D6, or strong inhibitors or inducers of all major CYP450 isozymes that cannot be stopped at least 7 days or 5 half-lives (whichever is longer) before starting treatment with ABC294640 and either replaced with another appropriate medication or not given for the duration of the clinical study. (A list of commonly used drugs that are sensitive substrates of CYP450 1A2, 3A4, 2C9, 2C19 or 2D6, or strong inhibitors or inducers of all major CYP450 isozymes with the half-life of each drug identified, is included as an Appendix C)
13. A history of CTC Grade 3 bleeding esophageal or gastric varices within the past 2 months. Prior variceal bleed is permitted if patient has undergone banding or sclerotherapy and there has been no evidence of bleeding for 2 months. Patients at risk for varices (based on the following: known history of esophageal or gastric varices; evidence of hepatic cirrhosis and/or portal hypertension including biopsy-proven cirrhosis, hypersplenism, or radiographic findings of varices) will be screened (using either esophagogastroduodenoscopy (EGD) or capsule endoscopy) for esophageal varices, unless such screening has been performed in the past two years from study entry and the patient is receiving medical treatment for prophylaxis of variceal bleeding, such as non-selective beta blockade. If varices are identified that require intervention (banding), patient will not be eligible until varices are adequately treated. Patients presenting with gastric varices will not be eligible for the study.
14. Patients who are currently taking Coumadin or Coumadin derivatives.
15. Patients who are currently participating in any other clinical trial of an investigational product.
16. History of organ transplantation.
17. Other primary malignancy within past 5 years except carcinoma in situ of the cervix or urinary bladder or non-melanoma skin cancer.
18. Any other mental incapacitation or psychiatric illness that would preclude study participation, as determined by the enrolling investigator.
19. Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
To assess objective response rate (per modified RECIST) of single agent ABC294640 in treatment of HCC | The primary endpoint is objective response rate (ORR) at 16 weeks defined according to modified RECIST criteria in second-line ABC294640 in patients with advanced HCC who have progressed on sorafenib.
  Radiographic Assessment will be completed up to 28 days prior to registration and every 8 weeks (+/- 7 days) following registration until disease progression or other (e.g.toxicity, patient decision, etc). The baseline radiographic assessment will include CT or MRI of the chest, abdomen and pelvis. Subsequent imaging will include only those body regions that include measureable index lesions per modified RECIST. Radiographic assessments will be completed every 8 weeks (+/- 7 days). In regards to the end of treatment visit, if the patient is taken off study and already has radiographic documentation of progressive disease, completing the radiographic assessment at the end of treatment visit is not required per study. If the patient is taken off study for other reasons such as toxicity or patient decision, it is strongly recommended that a radiographic assessment be obtained.

SECONDARY OUTCOMES:
To estimate the time to tumor progression (TTP) in HCC patients treated with ABC294640 | While on study, radiographic response will be documented every 8 weeks; after discontinuation, every 3 months for a maximum of 24 months after the last patient registered
  Patients who have not progressed by the end of the follow-up will have their TTP values censored.
To estimate the overall survival (OS) in HCC patients treated with ABC294640 | Time interval from initiation of study treatment to death due to any cause. All patients should be followed every 3 months for survival for a maximum of 24 months after the last patient has been registered to the trial.
  Survival times will be censored for patients lost to follow-up or still alive at the trial's termination.
To evaluate the pharmacokinetic behavior of ABC294640 in HCC patients [Peak Plasma Concentration (Cmax)] | From Cycle 1 Day 1 through to prior to dosing in Cycle 2 Day 1. (Each cycle is 28 days)
  Blood samples will be drawn. Plasma or PK analysis for ABC294640 will be collected on:
  * Cycle 1 (each cycle is 28 days) Day 1 prior to and at 2 and 8 hours post ABC294640 dosing
  * Prior to dosing on and at 2 hours post dose Cycle 1 Day 15
  * Prior to dosing on Cycle 2 Day 1.
To evaluate the pharmacokinetic behavior of ABC294640 in HCC patients [Area Under the drug concentration over time curve, (AUC)] | From Cycle 1 Day 1 through to prior to dosing in Cycle 2 Day 1. (Each cycle is 28 days)
  Blood samples will be drawn. Plasma or PK analysis for ABC294640 will be collected on:
  * Cycle 1 (each cycle is 28 days) Day 1 prior to and at 2 and 8 hours post ABC294640 dosing
  * Prior to dosing on and at 2 hours post dose Cycle 1 Day 15
  * Prior to dosing on Cycle 2 Day 1.
To describe the relationship between changes in marker levels of sphingolipids in peripheral blood in patients being given ABC294640 | Plasma samples for sphingolipid profiling will be drawn at baseline, on Cycle 1 Day 1 prior to and 8 hours post ABC dosing, and prior to dosing on Cycle 1 Day 15 and Cycle 2 Day 1, and within 1 hour prior to the pre- and post-treatment tumor biopsies.
  Scatterplots of percent change in target lesions versus change in marker levels will be constructed. Variable transformations will be considered as needed and Pearson or Spearman correlation coefficients will be constructed as appropriate. The sample size of 39 provides a minimum of 80% power to detect a correlation of at least ± 0.44 versus a null correlation of 0.
To explore the relationship between changes in c-Myc marker levels in peripheral blood mononuclear cells in patients being given ABC294640 | Peripheral Blood Mononuclear Cells (PBMC) for c-Myc will be collected within 1 hour prior to the pre- and post-treatment biopsies.
  Scatterplots of percent change in target lesions versus change in marker levels will be constructed. Variable transformations will be considered as needed and Pearson or Spearman correlation coefficients will be constructed as appropriate. The sample size of 39 provides a minimum of 80% power to detect a correlation of at least ± 0.44 versus a null correlation of 0.
To assess the relationship between changes in marker levels of sphingolipids in tumor tissue from patients being given ABC294640. | Tumor biopsies will be obtained within 28 days prior to Cycle 1 (each cycle is 28 days) Day 1, and again on Cycle 2 Day 1 (+/- 7 days), and will be assessed for tumor sphingolipid profile and tumor signaling proteins (c-Myc, pAKT, SK2).
  Scatterplots of percent change in target lesions versus change in marker levels will be constructed. Variable transformations will be considered as needed and Pearson or Spearman correlation coefficients will be constructed as appropriate. The sample size of 39 provides a minimum of 80% power to detect a correlation of at least ± 0.44 versus a null correlation of 0.
To assess the relationship between changes in c-myc marker levels in tumor tissue from patients being given ABC294640. | Tumor biopsies will be obtained within 28 days prior to Cycle 1 (each cycle is 28 days) Day 1, and again on Cycle 2 Day 1 (+/- 7 days), and will be assessed for tumor sphingolipid profile and tumor signaling proteins (c-Myc, pAKT, SK2).]
  Scatterplots of percent change in target lesions versus change in marker levels will be constructed. Variable transformations will be considered as needed and Pearson or Spearman correlation coefficients will be constructed as appropriate. The sample size of 39 provides a minimum of 80% power to detect a correlation of at least ± 0.44 versus a null correlation of 0.
Descriptive statistics of adverse events reported in all subjects treated with ABC294640 | The study period during which all AEs and SAEs must be reported begins after initiation of study treatment and ends 30 days following the last administration of study treatment.
  All AEs and SAEs whether volunteered by the subject, discovered by study personnel during questioning, or detected through physical examination, laboratory test, or other means will be reported appropriately. Each reported AE or SAE will be described by its duration (i.e., start and end dates), regulatory seriousness criteria if applicable, suspected relationship to the study, and actions taken. Adverse events will be coded by body system and summary of table with incidence rates of AEs will be generated. Severity, duration, investigator attributed relationship to study drug and adverse event outcomes will be reported.
Descriptive statistics of adverse events reported in subjects who discontinued study drug due to adverse events | The study period during which all AEs and SAEs must be reported begins after initiation of study treatment and ends 30 days following the last administration of study treatment.
  All AEs and SAEs whether volunteered by the subject, discovered by study personnel during questioning, or detected through physical examination, laboratory test, or other means will be reported appropriately. Each reported AE or SAE will be described by its duration (i.e., start and end dates), regulatory seriousness criteria if applicable, suspected relationship to the study, and actions taken. Adverse events will be coded by body system and summary of table with incidence rates of AEs will be generated. Severity, duration, investigator attributed relationship to study drug and adverse event outcomes will be reported.
Descriptive statistics of adverse events reported in subjects with adverse events related to study drug. | The study period during which all AEs and SAEs must be reported begins after initiation of study treatment and ends 30 days following the last administration of study treatment.
  All AEs and SAEs whether volunteered by the subject, discovered by study personnel during questioning, or detected through physical examination, laboratory test, or other means will be reported appropriately. Each reported AE or SAE will be described by its duration (i.e., start and end dates), regulatory seriousness criteria if applicable, suspected relationship to the study, and actions taken. Adverse events will be coded by body system and summary of table with incidence rates of AEs will be generated. Severity, duration, investigator attributed relationship to study drug and adverse event outcomes will be reported.
To assess the relationship between changes in immune cell subsets in peripheral blood from subjects being given ABC294640 | Blood will be drawn at baseline, on Cycle 1 Day 1 prior to and 8 hours post ABC294640 dosing, prior to dosing on Cycle 1 Day 15 and Cycle 2 Day 1, and within 1 hour prior to the pre-and post-treatment tumor biopsies.
  Scatterplots of percent change in target lesions versus change in immune cell subsets will be constructed. Variable transformations will be considered as needed and Pearson or Spearman correlation coefficients will be constructed as appropriated. The sample size of 39 provides a minimum of 80% power to detect a correlation of at least ± 0.44 versus a null correlation of 0.

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States